CLINICAL TRIAL: NCT04734912
Title: Evaluation of Transnasal Endoscopy During COVID-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Prof. Helmut Neumann, Principal Investigator, Johannes Gutenberg University Mainz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ETNE v1.0
Record Dates: First submitted 2021-01-13; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Endoscopy
Keywords: gastroscopy; transnasal; nursing
MeSH Terms: interventions — Gastroscopy

STUDY DESIGN:
Intervention Model Description: all patients with indication für gastroscopy in transnasal techique are included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastroscopy in transnasal technique (Other): All patients with indication for gastroscopy in transnasal techqiue are included.
  Interventions: Other: gastroscopy in transnasal techique

INTERVENTIONS:
Other: gastroscopy in transnasal techique — All patients with indication for gastroscopy in transnasal technique are included.

SUMMARY:
Patients who received the indication for endoscopic diagnostics using gastroscopy in transnasal technique will be included into the study. The examination is carried out in standard technique and is not influenced by the study. Following the examination, patient data is collected pseudonymously and a questionnaire is submitted to the patient.

DETAILED DESCRIPTION:
COVID-19 is transmitted, among other things, by a droplet infection. Conventional gastroscopy through the patient's mouth is therefore considered a high-risk examination for the medical and nursing staff. Alternatively, gastroscopy can also be performed through the patient's nose. An advantage here is that the aerosol formation is naturally significantly reduced and the patient usually does not need sedation, since in transnasal endoscopy no stranglehold occurs. Transnasal endoscopy therefore appears to us, especially during the COVID-19 pandemic, as a safe alternative to conventional gastroscopy.

Patients who received the indication for endoscopic diagnostics using gastroscopy in transnasal technique will be included into the study. The examination is carried out in standard technique and is not influenced by the study. Following the examination, patient data is collected pseudonymously and a questionnaire is sumbitted to the patient.

Only patients who have the indication for gastroscopy in transnasal technique are included. A specific risk to patients cannot be foreseen.This study does not interfere with diagnostics or therapy.

ELIGIBILITY:
Inclusion Criteria:

* Indication for transnasal endoscopy

Exclusion Criteria:

* pregnancy
* breast feeding
* contraindication to transnasal endoscopy
* pronounced blood clotting disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | after examination, about 15 minutes
  a questionnaire with 5 questions regarding the quality of the examination, technique and safety is presented to the patients

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Neumann, M.D. PhD, Principal Investigator — University Medical Center Mainz
Locations (1):
- University Hospital Mainz, Mainz, Rhenanie-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No
A publication of the results is planned.